CLINICAL TRIAL: NCT06105021
Title: Phase I Study of Autologous CD8+ and CD4+ Engineered T Cell Receptor T Cells in Subjects With Advanced or Metastatic Solid Tumor
Status: Active, not recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Affini-T Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: AFNT211-22-101
Record Dates: First submitted 2023-10-09; First posted 2023-10-27 (Actual); Last update posted 2025-07-30 (Actual); Status verified 2025-07

CONDITIONS: Pancreatic Ductal Adenocarcinoma; Non-Small Cell Lung Cancer; Colorectal Cancer; Solid Tumor; KRAS G12V
Keywords: PDAC; NSCLC; CRC; human leukocyte antigen-A; Kirsten rat sarcoma; HLA-A*11:01; KRAS; G12V; LDC; Lymphodepleting chemotherapy
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Colorectal Neoplasms; Syndactyly, Type I

STUDY DESIGN:
Intervention Model Description: This is a Phase I, FIH, multicenter, open-label study of AFNT-211 consisting of a dose escalation part and a dose expansion part. During dose escalation the optimal biological dose (OBD) will be determined as well as the recommended phase 2 dose (RP2D). Additional subjects will enroll in expansion cohorts treated at OBD/RP2D found in escalation.
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- Dose Escalation (Experimental): Subjects will be given a one-time infusion of AFNT-211 starting at dose level 1 and monitored for 28 days (DLT period). Each cohort will enroll 2-4 subjects at different dose levels for a total of 20 subjects in the escalation portion. The optimal biological dose and recommended phase 2 dose will be determined.
  Interventions: Drug: AFNT-211
- Dose Expansion: PDAC (Experimental): 20 subjects with pancreatic ductal adenocarcinoma will be given a one-time infusion of AFNT-211 at the optimal biological dose / recommended phase 2 dose determined in the escalation portion. Subjects will be monitored for safety for 28 days.
  Interventions: Drug: AFNT-211
- Dose Expansion: CRC (Experimental): 20 subjects with colorectal carcinoma will be given a one-time infusion of AFNT-211 at the optimal biological dose / recommended phase 2 dose determined in the escalation portion. Subjects will be monitored for safety for 28 days.
  Interventions: Drug: AFNT-211
- Dose Expansion: NSCLC (Experimental): 20 subjects with non-small cell cancer will be given a one-time infusion of AFNT-211 at the optimal biological dose / recommended phase 2 dose determined in the escalation portion. Subjects will be monitored for safety for 28 days.
  Interventions: Drug: AFNT-211
- Dose Expansion: Adv Solid Tumors (Experimental): 20 subjects with solid tumors will be given a one-time infusion of AFNT-211 at the optimal biological dose / recommended phase 2 dose determined in the escalation portion. Subjects will be monitored for safety for 28 days.
  Interventions: Drug: AFNT-211

INTERVENTIONS:
Drug: AFNT-211 — Engineered TCR T-Cell

SUMMARY:
This study is open to adult patients with solid tumors who have a KRAS G12V mutation. This mutation is often found in non-small cell lung cancer (NSCLC), colorectal cancer (CRC), pancreatic ductal adenocarcinoma (PDAC) and other cancers. The study is for patients whose cancer has spread through the body and for whom previous treatments were not successful or treatment does not exist. Patients must also be positive for HLA-A*11:01. The purpose of this study is to find the best dose of AFNT-211 that is safe and can shrink tumors in patients. AFNT-211 is an investigational therapy and this is the first time that AFNT-211 is being administered to patients. AFNT-211 is an autologous T cell product which means that it is made from a patient's own T cells. These cells are engineered and grown to recognize the KRAS G12V protein on the cell surface of cancer cells. AFNT-211 is infused into patients after a short course of lymphodepleting chemotherapy. Patients will frequently visit the study site. The doctors there will regularly check the size of the cancer and the patient's health. They will also take note of any unwanted effects. Patients may continue in this study for as long as they benefit from the treatment.

DETAILED DESCRIPTION:
AFNT-211 is a cellular therapy consisting of autologous CD4+ and CD8+ T cells engineered to express a human leukocyte antigen-A (HLA-A)*11:01-restricted Kirsten rat sarcoma (KRAS) G12V-specific transgenic T cell receptor (TCR), the wildtype CD8α/β coreceptor, and a FAS-41BB switch receptor. AFNT-211 is being developed by Affini-T Therapeutics, Inc. (hereafter, "the Sponsor") for the treatment of patients with malignant solid tumors. The primary purpose of this study is to assess the safety and tolerability of AFNT-211 in subjects who are HLA-A*11:01 positive with advanced or metastatic cancers that harbor a KRAS G12V mutation, as well as determine the optimal biological dose (OBD) and recommended Phase II dose (RP2D) of AFNT-211 in this population. This study will also evaluate the preliminary anti-tumor activity of AFNT-211.

ELIGIBILITY:
Key Inclusion Criteria:

1. Confirmed KRAS G12V mutational status and HLA-A*11:01 allele
2. Histologically confirmed advanced or metastatic, unresectable solid tumor
3. Progressed on or intolerant of at least one prior line of standard systemic therapy for the current malignancy.
4. Measurable disease per RECIST v1.1.
5. ECOG performance status 0-1
6. Adequate organ and bone marrow function

Key Exclusion Criteria:

1. Any systemic cytotoxic chemotherapy, investigational agents, or any anti-tumor drug from a previous treatment regimen or clinical study (including small molecules and I/O compounds) within 5 half-lives or 14 days of Screening, whichever is shorter.
2. Any prior gene therapy utilizing an integrating vector
3. Previous allogeneic stem cell transplantation or prior organ transplantation
4. History of treated primary immunodeficiency, autoimmune, or inflammatory disease including inflammatory bowel disease, systemic lupus erythematosus, rheumatoid arthritis, myasthenia gravis, or Grave's disease
5. Primary brain tumor
6. Untreated central nervous system (CNS) metastatic disease, leptomeningeal disease, or cord compression.
7. Uncontrolled active bacterial, viral, fungal, or mycobacterial infection
8. Pregnant or lactating subjects
9. Surgery or catheter-based interventions
10. Previously identified allergy, hypersensitivity, or known contraindication to cyclophosphamide, fludarabine, or any other agent associated with lymphodepleting chemotherapy (LDC) or AFNT-211 product
11. Uncontrolled significant intercurrent or recent illness
12. Diagnosis of another malignancy within 2 years prior to screening.
13. Seropositive for hepatitis B surface antigen (HBsAg) and/or hepatitis B core antibody (HBcAb)
14. Seropositive for hepatitis C antibody.
15. Known human immunodeficiency virus (HIV) infection

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2024-03-06 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2029-12 (Estimated)

PRIMARY OUTCOMES:
Determine the Optimal Biological Dose (OBD) | 60 months
  Quantify the desirability of a dose in terms of toxicity-efficacy tradeoff during the dose escalation portion of the study
Determine the Recommended Phase 2 Dose | 60 months
  This will be selected based on Bayesian optimal interval Phase I/II (BOIN12) design recommendation and the totality of benefit-risk evidence during dose escalation
Incidence of Treatment Emergent Adverse Events | 60 months
  The incidence of TEAEs will be used to determine safety and tolerability of AFNT-211
Incidence of Serious Adverse Events | 60 months
  The incidence of SAEs will be used to determine safety and tolerability of AFNT-211
Incidence of Dose Limiting Toxicities | 18 months
  The incidence of DLTs during Dose Escalation will be used to determine safety and tolerability of AFNT-211

SECONDARY OUTCOMES:
Overall Response Rate (ORR) | 60 months
  Percentage of subjects who achieved partial response (PR) or complete response (CR) as determined by Response Evaluation Criteria in Solid Tumors (RECIST) v1.1
Duration of Response (DOR) | 60 months
  Time from first documentation of response of PR or better to first documentation of disease progression or death from any cause, whichever occurs first.
Progression-free Survival (PFS) | 60 months
  From enrollment to first documentation of disease progression or death of any cause, whichever occurs first.
Time to Response (TTR) | 60 months
  Time from first AFNT-211 infusion to first documentation of PR or better.
Clinical Benefit Rate (CBR) | 60 months
  Percentage of subjects who have achieved PR or CR, or had stable disease (SD) for 6 months or more.
Overall Survival (OS) | 60 months
  From time of enrollment to death from any cause

CONTACTS AND LOCATIONS:
Locations (10):
- United States (10):
  - USC Norris Comprehensive, Los Angeles, California
  - University of California Los Angeles Department of Medicine, Los Angeles, California
  - Yale New Haven Hospital, New Haven, Connecticut
  - Laura & Isaac Perlmutter Cancer Center at NYU Langone Health, New York, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Providence Cancer Institute Franz Clinic, Portland, Oregon
  - Sarah Cannon Research Institute, Nashville, Tennessee
  - MD Anderson Cancer Center, Houston, Texas
  - Fred Hutchinson Cancer Center, Seattle, Washington
  - University of Wisconsin Carbone Cancer Center, Madison, Wisconsin

IPD SHARING:
Plan to Share IPD: No